CLINICAL TRIAL: NCT03030287
Title: A Phase 1b Study of OMP-305B83 Plus Weekly Paclitaxel in Subjects With Platinum Resistant Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: A Phase 1b Study of OMP-305B83 Plus Paclitaxel in Subjects With Ovarian, Peritoneal or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B83-002
Record Dates: First submitted 2017-01-13; First posted 2017-01-25 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Cancer Ovaries; Cancer Peritoneal; Cancer, Fallopian Tube
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — navicixizumab; Antibodies, Bispecific; Paclitaxel

ARMS (1):
- OMP-305B83 plus paclitaxel (Experimental)
  Interventions: Drug: OMP-305B83; Drug: Paclitaxel

INTERVENTIONS:
Drug: OMP-305B83 — intravenous (in the vein) infusion
  Other Names: bispecific monoclonal antibody
Drug: Paclitaxel — administered intravenously

SUMMARY:
The purpose of this study is to test the efficacy and safety of an experimental drug, OMP-305B83, when given in combination with paclitaxel. OMP-305B83 is a humanized monoclonal antibody and was developed to target cancer stem cells. Based on preclinical studies, it is believed that OMP-305B83 may block the growth of cancer stem cells and may also impair the productive growth of new blood vessels, which tumors need to grow and spread.

DETAILED DESCRIPTION:
This is an open-label, Phase 1b dose escalation and expansion study of OMP-305B83 plus paclitaxel designed to evaluate the safety, efficacy and pharmacokinetics of OMP-305B83 in combination with paclitaxel in patients with platinum resistant ovarian, primary peritoneal or fallopian tube cancer. This study consists of a screening period, a treatment period and a post-treatment follow up period in which patients will be followed for survival for approximately 12 months. Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase.

Approximately 30 patients will be enrolled in this study at approximately 5 study centers in the United States (U.S)..

ELIGIBILITY:
Inclusion Criteria:

1. Platinum resistant Grade 2 or 3 ovarian, primary peritoneal or fallopian tube cancer
2. Measureable disease per response evaluation criteria (RECIST) v1.1
3. Prior bevacizumab
4. Age > or = 21 years
5. Adequate organ and marrow function
6. For women of childbearing potential and men with partners of childbearing potential, agreement (by patient and/or partner) to use two effective forms of contraception from study entry through at least 6 months after the termination visit.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Treatment with any anti-cancer therapy, including radiotherapy, chemotherapy, biologic therapy. Prior therapy with weekly paclitaxel for recurrent disease, unless administered more than 2 years prior to enrollment, unless part of an upfront treatment strategy.
2. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, clinical signs or symptoms of gastrointestinaI obstruction or other known clinically signification gastrointestinal disease.
3. Subjects with brain metastases
4. Subjects with leptomeningial disease or neoplasms in the last 5 years
5. Blood pressure >140/80
6. Significant intercurrent illness that will limit the patient's ability to participate in the study
7. Subjects with known metastases that are currently involving the lumen of the gastrointestinal tract.
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment, or anticipation of need for major surgical procedure during the course of the study
9. Pregnant or nursing women
10. New York Heart Association Classification II, III, or IV
11. Inability to comply with study and follow up procedure

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-12; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLT) | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-28).
  The maximum tolerated dose (MTD) or maximum administered dose (MAD) will be determined in subjects treated with OMP-305B83 in combination with Paclitaxel

SECONDARY OUTCOMES:
Safety of OMP-30B583 in combination with Paclitaxel will be assessed by adverse event monitoring, physical exams, vital signs, clinical laboratory testing, ECGs, echocardiograms, anti-OMP-305B83 testing, and subject interview on an ongoing basis. | Through study completion, an average of 6 months
To assess Immunogenicity (in terms of formation of anti-drug antibod(ies) against OMP-305B83 in percentage of subjects) of OMP-305B83 in combination with Paclitaxel | Through study completion, an average of 6 months
Response Rate assessed by RECIST criteria 1.1 | At 56 day intervals while on treatment, through study completion, an average of 6 months
Response Rate assessed by CA-125 criteria | At 28 day intervals while on treatment, through study completion, an average of 6 months
Progression Free Survival | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Inc. (Moffitt Cancer Center), Tampa, Florida
  - Levine Cancer Institute, Charlotte, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - The University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Fu S, Corr BR, Culm-Merdek K, Mockbee C, Youssoufian H, Stagg R, Naumann RW, Wenham RM, Rosengarten RD, Benjamin L, Hamilton EP, Moore KN. Phase Ib Study of Navicixizumab Plus Paclitaxel in Patients With Platinum-Resistant Ovarian, Primary Peritoneal, or Fallopian Tube Cancer. J Clin Oncol. 2022 Aug 10;40(23):2568-2577. doi: 10.1200/JCO.21.01801. Epub 2022 Apr 19. PMID 35439029